CLINICAL TRIAL: NCT06830798
Title: A Phase 3, Double-blind, Randomized, Placebo-controlled, Multicenter Study to Evaluate the Efficacy and Safety of Ravulizumab Administered Intravenously in Adult Participants at High Risk of Delayed Graft Function After Kidney Transplantation
Brief Title: Double-blind, Randomized, Placebo-controlled, Multicenter Study to Evaluate the Efficacy and Safety of Ravulizumab Administered Intravenously in Adult Participants at High Risk of Delayed Graft Function After Kidney Transplantation
Acronym: AWAKE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D928EC00001; 2024-517568-48 (EudraCT Number)
Record Dates: First submitted 2025-02-10; First posted 2025-02-17 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Delayed Graft Function; DGF; Kidney Transplant
Keywords: Delayed Graft Function; DGF; Kidney Transplant; Ravulizumab
MeSH Terms: conditions — Delayed Graft Function | interventions — ravulizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ravulizumab (Experimental): Participants will receive an IV dose of ravulizumab.
  Interventions: Drug: Ravulizumab
- Placebo (Placebo Comparator): Participants will receive an IV dose of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ravulizumab — Participants will receive ravulizumab via intravenous (IV) infusion.
  Arms: Ravulizumab
Drug: Placebo — Participants will receive placebo via intravenous (IV) infusion.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to demonstrate the efficacy of ravulizumab vs placebo in reducing the severity of DGF as measured by time to freedom from dialysis in adult participants who are at high risk of DGF after undergoing transplant of deceased donor kidney.

DETAILED DESCRIPTION:
AWAKE is a multicenter, prospective study to evaluate the safety and efficacy of ravulizumab in reducing delayed graft function (DGF) in kidney transplant recipients at high risk for DGF. Eligible participants will be randomized in a 1:1 ratio to receive either ravulizumab or placebo intravenously.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age at the time of signing the informed consent
* Diagnosed with Dialysis-dependent End-Stage Kidney Disease (ESKD)
* A candidate for kidney transplant from:

  1. Donation after Circulatory Death (DCD) donor
  2. High-risk Donation after Brain Death (DBD) donor

Exclusion Criteria:

* Is to receive a kidney from a donor with category I,II,IV and V Maastricht Classification
* Diagnosed with Acute Kidney Injury (AKI) of Stage 3 severity according to the Kidney Disease: Improving Global Outcomes (KDIGO) guidelines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2028-02-04 (Estimated); Study Completion 2028-11-06 (Estimated)

PRIMARY OUTCOMES:
Time to Freedom from Dialysis | Through 90 days post-transplant

SECONDARY OUTCOMES:
DGF Incidence | Up to 7 days post-transplant
Number of Dialysis Sessions | Through 90 days post-transplant
Time to Occurrence of eGFR reaching 30 mL/min/1.73 m2 | Through 90 days post-transplant

CONTACTS AND LOCATIONS:
Locations (105):
- United States (29):
  - Research Site, Phoenix, Arizona
  - Research Site, Los Angeles, California
  - Research Site, San Francisco, California
  - Research Site, Stanford, California
  - Research Site, New Haven, Connecticut
  - Research Site, Jacksonville, Florida
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Fairway, Kansas
  - Research Site, Lexington, Kentucky
  - Research Site, Kenner, Louisiana
  - Research Site, Ann Arbor, Michigan
  - Research Site, Detroit, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Omaha, Nebraska
  - Research Site, Livingston, New Jersey
  - Research Site, New York, New York
  - Research Site, Durham, North Carolina
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Greenville, South Carolina
  - Research Site, Nashville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Charlottesville, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Seattle, Washington
  - Research Site, Milwaukee, Wisconsin
- Argentina (3):
  - Research Site, Buenos Aires
  - Research Site, Capital Federal
  - Research Site, Córdoba
- Australia (4):
  - Research Site, Adelaide
  - Research Site, Brisbane
  - Research Site, Camperdown
  - Research Site, Murdoch
- Austria (2):
  - Research Site, Innsbruck
  - Research Site, Vienna
- Brazil (9):
  - Research Site, Belo Horizonte
  - Research Site, Botucatu
  - Research Site, Campinas
  - Research Site, Fortaleza
  - Research Site, Porto Alegre
  - Research Site, Recife
  - Research Site, Rio de Janeiro
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
- Canada (3):
  - Research Site, Edmonton, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Toronto, Ontario
- China (8):
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Hengyang
  - Research Site, Nanning
  - Research Site, Shenzhen
  - Research Site, Taiyuan
  - Research Site, Tianjin
  - Research Site, Zhengzhou
- Czechia (3):
  - Research Site, Hradec Kralova
  - Research Site, Ostrava
  - Research Site, Prague
- France (7):
  - Research Site, Créteil
  - Research Site, La Rochelle
  - Research Site, La Tronche
  - Research Site, Montpellier
  - Research Site, Nantes
  - Research Site, Paris
  - Research Site, Toulouse
- Germany (5):
  - Research Site, Berlin
  - Research Site, Erlangen
  - Research Site, Lübeck
  - Research Site, Mainz Am Rhein
  - Research Site, Münster
- Italy (5):
  - Research Site, Bologna
  - Research Site, Milan
  - Research Site, Padua
  - Research Site, Parma
  - Research Site, Torino
- Japan (2):
  - Research Site, Kyoto
  - Research Site, Suita-shi
- Poland (4):
  - Research Site, Bydgoszcz
  - Research Site, Gdansk
  - Research Site, Poznan
  - Research Site, Warsaw
- Portugal (2):
  - Research Site, Lisbon
  - Research Site, Porto
- South Korea (2):
  - Research Site, Gyeonggi-do
  - Research Site, Seoul
- Spain (10):
  - Research Site, Badajoz
  - Research Site, Barakaldo
  - Research Site, Barcelona
  - Research Site, Cadiz
  - Research Site, Córdoba
  - Research Site, Granada
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Valencia
  - Research Site, Zaragoza
- Taiwan (4):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Taipei
  - Research Site, Taoyuan District
- United Kingdom (3):
  - Research Site, Leeds
  - Research Site, London
  - Research Site, Woodville South

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.
Supporting Information: Study Protocol, SAP, CSR